CLINICAL TRIAL: NCT06130241
Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Initially Node Positive Breast Cancer Patients, Could it Omit Axillary Dissection ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hosny Mahmoud, Resident doctor at general surgery department in Assuit university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sentinel L.N in breast cancer
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Sentinel Lymph Node

STUDY DESIGN:
Intervention Model Description: female with breast cancer and malignant axillary lymphnodes who underwent neoadjuvant chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- female with breast cancer and positive axillary lymphnodes (Other): female patients with breast cancer with initially positive axillary lymphnodes who underwent neoadjuvant chemotherapy
  Interventions: Procedure: sentinle lymphnode biopsy

INTERVENTIONS:
Procedure: sentinle lymphnode biopsy — intraoperative sentinle lymphnode biopsy

SUMMARY:
The aim of this study is to determine the accuracy and safety of SLNB after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women. The morbidity and mortality of breast cancer are much higher than those observed with other female cancers . The incidence of breast cancer increases with age.

Approximately 1.7 million new cases are estimated to occur worldwide, and mortality is increasing in developing countries, primarily because the disease is not diagnosed until it is in an advanced stage

Neoadjuvant chemotherapy (NACT) is considered the standard of care for the anagement of locally advanced breast cancer and although this treatment has historically been reserved for those with inoperable breast cancer now is increasingly being used for women with earlier stage disease.

. Encouraging results obtained with neoadjuvant chemotherapy in have resulted in clinicians using preoperative chemotherapy for patients with smaller tumors.

Neoadjuvant chemotherapy (NACT) could reduce surgical morbidity of the breast and axilla. By down staging of the tumor, NACT can convert patients who are candidates for mastectomy to breast-conserving surgery (BCS) candidates .

Furthermore, it has potential to reduce excision volumes in patients with large tumors who are already candidates for BCS. Another surgical advantage is down staging of the axilla so that axillary lymph node dissection can be avoided .

In the treatment of breast cancer, sentinel lymph node biopsy (SLNB) has replaced axillary lymph node dissection (ALND) as the staging procedure for patients with clinically node-negative disease. It provides accurate assessment of histological nodal status, guides additional therapies and is associated with less morbidity than ALND. Historically, patients who were clinically node-negative would undergo SLNB, whereas patients who were node-positive underwent ALND. SLNB in the neoadjuvant setting has become a topic of debate. Unfortunately, the reliability of SLNB after NAC remains questionable. Chemotherapy causes fibrosis, fat necrosis and granulation tissue formation, which alters lymphatic drainage patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with operable breast cancer who had node-positive disease at presentation and pathological confirmation with either FNA or core biopsy
2. Female Patient aged from 18 to 60 years old
3. Patients who are fit for general anesthesia.
4. Patient who agree to provide short term outcome data and agree to provide contact information to provide contact information.

Exclusion Criteria:

1. Stage 4 breast cancer
2. Patient has no clinical response to NACT
3. Patients who are contraindicated for radiotherapy
4. Pregnant patients in first trimester
5. Patient with inflammatory carcinoma

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients with breast cancer
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Initially Node Positive Breast Cancer Patients, Could it Omit Axillary Dissection? | Two year
  To evaluate the accuracy and safety of SLNB after neoadjuvant chemotherapy by 2 years follow up patients for recurrence clinically and radiologically by ultrasonography on axilla after one and two years .

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud thabet, Assistant lecture, Study Director — Assiut University; negm eldein abulnaga, lecturer of general surgery, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hery C, Ferlay J, Boniol M, Autier P. Changes in breast cancer incidence and mortality in middle-aged and elderly women in 28 countries with Caucasian majority populations. Ann Oncol. 2008 May;19(5):1009-18. doi: 10.1093/annonc/mdm593. Epub 2008 Feb 21. PMID 18296422
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Mieog JS, van der Hage JA, van de Velde CJ. Preoperative chemotherapy for women with operable breast cancer. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD005002. doi: 10.1002/14651858.CD005002.pub2. PMID 17443564
- [Result] Cleries R, Rooney RM, Vilardell M, Espinas JA, Dyba T, Borras JM. Assessing predicted age-specific breast cancer mortality rates in 27 European countries by 2020. Clin Transl Oncol. 2018 Mar;20(3):313-321. doi: 10.1007/s12094-017-1718-y. Epub 2017 Jul 19. PMID 28726040